CLINICAL TRIAL: NCT03392181
Title: PET/MRI for the Staging of Newly Diagnosed Prostate Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Edward Schaeffer, Chair, Department of Urology, Program of Director for GU Oncology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NU 17U12; STU00205957 (Other: Northwestern IRB); NCI-2018-00059 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-DCFPyL (Experimental)
  Interventions: Drug: 18F-DCFPyL

INTERVENTIONS:
Drug: 18F-DCFPyL — To determine whether PET/MR utilizing PYL improves pre-operative staging of prostate cancer prior to radical prostatectomy compared to MRI alone.

SUMMARY:
The purpose of this study is to gain understanding of how PET-MR (positron emission tomography-magnetic resonance imaging) using the substance 18F-DCFPyL (PyL) may help in diagnosing prostate cancer and in determining the stage of prostate cancer before surgery.

ELIGIBILITY:
Inclusion Criteria

* Patients must have a biopsy-proven diagnosis of high risk, very high risk, or locally advanced prostate cancer
* Patients must have a diagnosis of high risk, very high risk, or locally advanced prostate cancer per NCCN Guidelines (T3-T4 disease)
* Patients are healthy enough to be deemed surgical candidates with an ECOG performance status of 0-2
* Patients must be age ≥ 18 years
* Patients must agree to use adequate contraception (e.g. barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days following completion of the imaging
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria

* Patients who have contraindications to MRI (i.e. pacemakers, aneurysm clips or shaped fragments)
* Patients who are claustrophobic will be required to take an anti-anxiety medication prescribed by their physician one hour prior to the scan
* Patients may not be receiving any other treatments or investigational agents
* Patients with a GFR <30mL/min are ineligible to receive intravenous contrast per standard MR exclusion criteria
* Patients not interested in pursuing surgical intervention for their disease (i.e. refusing treatment or requesting radiation oncology referral)
* Patients who have received androgen deprivation therapy or prior surgery for prostate cancer
* Patients who report taking multivitamins and/or folate supplements on the day of the scan

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-06-08 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
PET/MR versus mp-MRI for the Staging of Newly Diagnosed Prostate Cancer | 5 years
  To determine if PSMA-Targeted PET/MRI improves pre-operative staging of prostate cancer prior to radical prostatectomy compared to MRI alone.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Schaeffer, MD/PhD, Principal Investigator — Chair, Department of Urology
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li EV, Schaeffer EM, Ramesh Kumar SKS, Zhou R, Yang XJ, Mana-Ay M, Vescovo M, Ho A, Keeter MK, Carr J, Casalino D, Kocherginsky M, Patel HD, Ross AE, Savas H. Utility of 18F-DCFPyL PET for local staging for high or very high risk prostate cancer for patients undergoing radical prostatectomy. Eur J Nucl Med Mol Imaging. 2025 Jun;52(7):2335-2342. doi: 10.1007/s00259-025-07133-1. Epub 2025 Feb 10. PMID 39928105